CLINICAL TRIAL: NCT02426528
Title: UR.CULT.HEA - URban Environment, CULTural Social Use of Space and HEAlth / Well-being Effect on Population: Study Protocol for a Cluster Randomized Trial
Brief Title: R.CULT.HEA - URban Environment, CULTural Social Use of Space and HEAlth / Well-being Effect on Population
Acronym: URCULTHEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Giorgio Tavano Blessi, Postdoctoral fellow, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UBologna
Record Dates: First submitted 2015-04-01; First posted 2015-04-27 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Personal Satisfaction; Health Behavior
MeSH Terms: conditions — Personal Satisfaction; Health Behavior | interventions — Culture Techniques

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cultural and Social exposure A (Experimental): Cultural and Social exposure
  Interventions: Other: Cultural and Social exposure
- Cultural and Social exposure B (No Intervention): Non Intervention (Control Group)

INTERVENTIONS:
Other: Cultural and Social exposure — The intervention protocol will consist of 24 months of guided exposure and participation in social and cultural activities undertaken in the "Casa del Popolo". The participant will be asked to register for a specific type of event (fine arts, performing arts, and social and volunteering activities), duration and date in order that this information can be supplied for further evaluation. Control group participants will be asked to carry on their lives normally and maintain regular cultural and social activity throughout the duration of the study. At twelve months from the beginning of the observation participants of both groups will be checked (intermediate phase).
  Arms: Cultural and Social exposure A

SUMMARY:
This cluster randomized trial will test the affect of individual participation in culturally- and socially-related activities on health and well-being, in comparison also with the classic individual determinant, in relation to urban renovation schemes. Investigators will using a questionnaire based on several areas such as individual psychological well-being (PGWBI), individual happiness positioning (Keyes Scale) and health status perception (SF-12 Health Survey). Secondary outcomes will be related to social capital density (relationships and trust), culture (participation) and religion. The survey will be undertaken in a mid-size Italian metropolitan area, namely the Metropolitan City of Bologna.

ELIGIBILITY:
Inclusion Criteria:

* Gender: men and women;
* Age range between 18 and 75 years old;
* Residency: in an area of 2 square kilometers surrounding the Casa del Popolo

Exclusion Criteria:

* participants no having the previous features

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 625 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
PGWBI (The Psychological General Well-Being Index) | after 24 months (end of study)
  This is a self-administrated test with 22 items that assesses the subjective perception of psychological well-being. It has been divided into 6 categories: anxiety, depression, self-control, positivity, well-being, and health and vitality

SECONDARY OUTCOMES:
MHC-SF (Mental Health Continuum - Long Form MHC-LF) | after 24 months (end of study)
  This is a self-administered form and represents the short version (14 items) of the Mental Health Continuum - Long Form MHC-LF (12), the original forty-item instrument. As for the long form, the short one has been designed to measure emotional, psychological and social well-being described by the two-continuum model of positive health (10). Within this framework, participants can be identified as flourishing, languishing or enjoying moderate mental health; in other words the aim is to assess positive or negative mental health as a function of emotional, psychological, and social well-being
SF-12 Health Survey | after 24 months (end of study)
  This is a self-administered test that assesses global health status but from the subjective point of view. It has been divided into two principal subscales: The Physical Component Summary (PCS) and the Mental Component Summary (MCS). In particular, it allows us to assess concepts involving health, physical functions, pain, general health, vitality, social functioning, emotional functioning and mental health